CLINICAL TRIAL: NCT07169747
Title: The Therapeutic Potential of Psilocybin in Anorexia Nervosa in Young Adults
Brief Title: Safety, Therapeutic Potential, and Mechanisms of Two Psilocybin Doses, Administered With Psychological Support in Young Adults With Anorexia Nervosa
Acronym: psiAN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Sten Theanders fond (Unknown); Lions Forskningsfond Skåne (Unknown); NorrskenMind (Unknown)
Responsible Party: Principal Investigator, Pouya Movahed Rad, Associate Professor and Senior Consultant in Psychiatry, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-515163-63-00; 2024-515163-63-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-21; First posted 2025-09-12 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Anorexia Nervosa
Keywords: Psilocybin; Anorexia Nervosa; Young adults; fMRI; BDNF; Adolescents
MeSH Terms: conditions — Anorexia Nervosa | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: If the psilocybin treatment is determined to be safe, tolerable and preliminarly effective, participants in the control group will have the option to swith to psilocybin treatment (while maintaining their usual specialized care). This will be offered after 6 months post-baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psilocybin with Psychological Support (Active Comparator): This arm will receive two separate doses of psilocybin 25 mg administered four weeks apart, with psychological support, along side treatment as usual. The psychological support includes preparation sessions before, support during, and integration sessions after psilocybin intake.
  Interventions: Drug: Psilocybin
- Treatment as Usual (No Intervention): This arm will receive treatment as usual which includes specialised care offered in an eating disorder unit in Region Skåne, Sweden. If the active treatment arm is determined to be safe, tolerable, and preliminarily effective during the follow-up assessment at 6 months, participants in the control group will have the option to switch to the active treatment while maintaining their usual specialised care.

INTERVENTIONS:
Drug: Psilocybin — The intervention consists of two oral doses of 25 mg synthetic psilocybin administered in a controlled clinical setting, combined with psychological support. The psychological support includes preparatory sessions prior to psilocybin administration, support during the drug experience and integration sessions following each dosing session.
  Arms: Psilocybin with Psychological Support

SUMMARY:
The goal of this clinical trial is to learn if psilocybin, given with psychological support, is safe and helps treat anorexia nervosa in young adults. Anorexia nervosa is a serious eating disorder that currently has no approved medicine. Psilocybin is a psychedelic substance that may help the brain form new connections, which could make it easier for people with anorexia nervosa to develop healthier ways of thinking.

The main questions this study aims to answer are:

* Is psilocybin with psychological support safe and well-tolerated?
* Does psilocybin with psychological support help lower symptoms of anorexia nervosa?
* How might psilocybin work in the brain to support recovery from anorexia?

This study will compare psilocybin with psychological support to Treatment as Usual (TAU). Participants in the study will be randomly placed into one of the two groups. There will be 40 patients with anorexia nervosa included, 20 per group. TAU includes the standard care people receive for anorexia nervosa in a specialized eating disorder clinic in Region Skåne, Sweden.

Participants will:

* Be between 16 and 35 years old and have anorexia nervosa
* Take psilocybin (25 mg) by mouth two times, four weeks apart
* Receive psychological support before, during, and after each dosing session (including preparation and integration sessions)
* Complete questionnaires, have brain scans (magnetic resonance imaging) and blood tests to learn more about how psilocybin may work
* Share their personal experiences as part of a qualitative interview

This study hopes to learn if psilocybin, when given with the right support, can be a helpful and safe option for people living with anorexia nervosa.

DETAILED DESCRIPTION:
Background and Rationale Anorexia Nervosa (AN) is one of the most lethal psychiatric disorders, with mortality rates approximately five times higher than that of the general population. AN affects multiple organ systems due to severe weight loss and malnutrition and hence leads to a substantial decline in health-related quality of life. While psychotherapies have shown partial efficacy, data suggest that only 46% of patients recover within four years, and 20% remain chronically ill. Relapse rates exceed 50% among those who recover, underscoring the need for more effective treatments. Research suggests that several psychological factors, such as challenges in regulating emotions, black-and-white thinking, mental rigidity, and a limited capacity for mentalization may contribute to the persistence of severe, chronic anorexia nervosa. The age of onset for AN typically shows a bimodal distribution, peaking at 14 and 18 years of age, motivating the design of including patients as young as 16 years old in this study.

Psilocybin, a serotonergic psychedelic compound, primarily acts as an agonist of the 5-HT2A receptor, inducing profound effects on cognition, emotion, perception, and self-awareness. Although research on psilocybin remains limited, clinical trials across psychiatric disorders suggest its potential therapeutic benefit. For example personality changes such as increased openness, have been observed to persist up to a year following a single high dose. The inclusion of 16-17-year-olds in this study is particularly novel, as research on psychedelic therapy in adolescents and young adults remains scarce.

Emerging evidence highlights how psychedelics may benefit AN patients, such as enhanced serotonin signaling and cognitive flexibility. The ability of psychedelics to foster cognitive flexibility, a well-documented phenomenon, is considered a key factor in therapeutic processes. This is especially relevant for AN, where rigid thinking and behavior contribute to treatment resistance. One pilot study demonstrated that a 25 mg psilocybin dose, combined with psychological support, was well-tolerated by female AN patients with a body mass index (BMI) >16. The study reported significant reductions in eating disorder symptoms at one month post-treatment, with only mild and transient adverse events.

Recent studies indicate that psilocybin induces significant changes in brain function and network organization across key regions. Notably, psilocybin disrupts connectivity in the default mode network by causing desynchronization across spatial scales. These findings suggest a neurobiological basis for psilocybin´s therapeutic effect. However, further research is needed to elucidate long-term effects, particularly in clinical context. Functional magnetic resonance imaging (fMRI) has demonstrated utility in detecting neuronal abnormalities in AN. This study's use of fMRI before and after psilocybin treatment will provide critical insights into the neurobiological impacts of psilocybin on AN.

Brain-Derived Neurotrophic Factor (BDNF) is a protein that plays a crucial role in neuroplasticity. Preclinical studies show that psilocybin promotes neuritogenesis and synaptic plasticity, potentially via increased cortical BDNF expression. Given that individuals with AN exhibit reduced serum BDNF levels, this study will assess changes in BDNF pre- and post-treatment to elucidate psilocybin's impact on neurobiological mechanisms. These insights may advance treatment optimization and efficacy predictions for AN patients.

Study Objectives Primary Objective is to assess the safety and tolerability of psilocybin 25 mg in young adults (16-35 years old) with anorexia nervosa. Secondary objectives include evaluating the efficacy of psilocybin with psychological support in reducing AN symptom compared to treatment as usual (TAU), investigate potential mechanisms of action through self-report questionnaires, neuroimaging and BDNF analysis, and conduct qualitative analysis of subjective experiences.

Trial Design and Procedures

This is a phase II, open-label, randomized controlled trial with two arms:

1. Active treatment arm; Two dosing sessions with psilocybin 25mg with psychological support alongside TAU.
2. Active comparator control arm; TAU only. The study will include 40 participants, 20 in each group. If the active treatment arm is determined to be safe, tolerable, and preliminarily effective during the follow-up assessment, participants in the control group will have the option to switch to the active treatment while maintaining their usual specialized care. The switch to psilocybin treatment will follow the same preparation, dosing, and integration protocols as outlined for the intervention group.

   This design minimizes ethical concerns regarding withholding a potentially effective treatment. Participants will be randomly assigned (1:1) to either the intervention or control group. Block randomization stratified by age group (16-18 and 19-35 years) will ensure balanced representation.

   Given the small sample size of 40 participants (20 per group), the statistical power to detect between-group differences is inherently limited, irrespective of blinding. As such, the trial is appropriately designed as a pilot study, with a primary focus on assessing safety, feasibility, and tolerability. To enhance interpretation, qualitative and neurobiological measures are also included. A formal power calculation was not conducted, in line with the exploratory nature of the study. The sample size was determined based on practical feasibility and aligns with current recommendations for early-phase trials of novel interventions. A post-hoc power analysis will be conducted to evaluate whether the sample size was sufficient to detect clinically meaningful changes in the primary outcomes.

   Details on location and Data Collection Methods All procedures will be conducted at the University Hospital for Psychiatry, Baravägen 1, Lund, except the fMRI assessments which are performed at the The National 7 Tesla (7T) Facility in Lund. All assessments will be carried out by qualified personnel appointed by the principal investigator, including medical doctors, nurses, and psychologists. The National 7T Facility will appoint qualified personnel for fMRI assessment. The duration of the entire trial is from the first screening of the first patient to the last follow up of the last patient. For each patient participant, the duration of the trial is from the screening to the last follow up at week 52 (12 month). Patient rehospitalization and additional interventions data are collected in patient journal registers.

   Screening Phase Screening includes psychiatric and medical history, inclusion/exclusion criteria assessment, safety blood tests (glucose, liver, kidney), electrocardiogram (ECG), informed consent (with a 2-week consideration period), pregnancy test and urine toxicology (U-tox). The time from screening to the first psilocybin dose must not exceed 8 weeks, regardless of washout status. Potential participants will be screened by a psychiatric clinician appointed by the principal investigator to ensure eligibility and understanding of the study requirements.

   Preparation Phase Preparation Session 1 (Week -1): Psychoeducation about psilocybin, breathing and relaxation techniques, rapport-building with therapists, and discussion of expectations and concerns.

   Preparation Session 2 & Baseline Assessment (Week 0): Conducted 7-10 days after Preparation 1, and 2-3 days before psilocybin dosing. Includes full baseline assessments (list provided as attachment to protocol:
   * Expectation of Treatment Scale (ETS-BF)
   * Readiness and Motivation Questionnaire (RMQ)
   * General Change Mechanisms Questionnaire (GCMQ)
   * Patient Health Questionnaire (PHQ-9)
   * Generalized Anxiety Disorder scale (GAD-7)
   * Eating Disorder Examination Questionnaire (EDE-Q )
   * Columbia-Suicide Severity Rating Scale (C-SSRS)
   * Brief Psychiatric Rating Scale - Extended (BPRS+)
   * Life Satisfaction Scale (LS)
   * Positive and Negative Affect Schedule (PANAS)
   * Harmony in Life Scale (HILS)
   * Ten Item Personality Inventory (TIPI)
   * Honesty-Humility Scale (HH) Vital signs, ECG, fasting glucose, urine drug screening, fMRI, BMI and blood sampling for BDNF and safety labs are also conducted.

   Dosing and Integration Phase Dosing Session 1 (Week 0): Psilocybin 25 mg under therapeutic support with ECG and blood pressure/pulse monitoring.

   Integration Session 1 (Day after Dosing 1): Reflection, fMRI, blood sampling (including glucose, liver, kidney, BDNF), and reassessments with RMQ, GCMQ, PHQ-9, GAD-7, C-SSRS, BPRS+, LS, PANAS, HILS, TIPI, ECG and blood pressure/pulse. Psychedelic Experience related scales; Altered States of Consciousness Rating Scale (5D-ASC), Mystical Experience Questionnaire (MEQ-4), Meaningful Life Experience Rating (MLE).

   Integration Session 2 (Week 1): Continued psychological integration support.

   Integration Session 3 (Week 2-3): Summary of first dosing experience and preparation for second dosing.

   Dosing Session 2 (Week 4): Second psilocybin 25 mg administration under identical conditions as first dosing session.

   Integration Session 4 (Day after Dosing 2): Reflection, blood sampling (including glucose, liver, kidney, BDNF), and reassessments with RMQ, GCMQ, PHQ-9, GAD-7, C-SSRS, BPRS+, LS, PANAS, HILS, TIPI, ECG and blood pressure/pulse. Psychedelic Experience related scales; Altered States of Consciousness Rating Scale (5D-ASC), Mystical Experience Questionnaire (MEQ-4), Meaningful Life Experience Rating (MLE).

   Integration Session 5 (Week 5-6): Final integration session and preparation for long-term follow-up.

   Primary Endpoint (Week 8)

   Includes full safety and outcome evaluations:
   * fMRI
   * blood sampling (including glucose, liver, kidney, glucose, BDNF)
   * Vital signs, ECG, U-tox
   * BMI
   * Adverse Event/Serious Adverse Event (AE/SAE) monitoring
   * Readiness and Motivation Questionnaire (RMQ)
   * General Change Mechanisms Questionnaire (GCMQ)
   * Patient Health Questionnaire (PHQ-9)
   * Generalized Anxiety Disorder scale (GAD-7)
   * Eating Disorder Examination Questionnaire (EDE-Q )
   * Columbia-Suicide Severity Rating Scale (C-SSRS)
   * Brief Psychiatric Rating Scale - Extended (BPRS+)
   * Life Satisfaction Scale (LS)
   * Positive and Negative Affect Schedule (PANAS)
   * Harmony in Life Scale (HILS)
   * Ten Item Personality Inventory (TIPI)
   * Honesty-Humility Scale (HH)

   Intensive Follow-Up Phase (Week 8-24)

   Follow-up visits at Week 12, 16, and 20 include:
   * Eating Disorder Examination Questionnaire (EDE-Q )
   * Columbia-Suicide Severity Rating Scale (C-SSRS)
   * Brief Psychiatric Rating Scale - Extended (BPRS+)
   * AE/SAE monitoring
   * BMI, blood pressure, ECG
   * Fasting glucose, U-tox

     6-Month Follow-Up (Week 24)

   Same as primary endpoint assessments, including:
   * blood sampling (including glucose, liver, kidney, BDNF)
   * Vital signs, ECG, U-tox
   * BMI
   * AE/SAE monitoring
   * Readiness and Motivation Questionnaire (RMQ)
   * General Change Mechanisms Questionnaire (GCMQ)
   * Patient Health Questionnaire (PHQ-9)
   * Generalized Anxiety Disorder scale (GAD-7)
   * Eating Disorder Examination Questionnaire (EDE-Q )
   * Columbia-Suicide Severity Rating Scale (C-SSRS)
   * Brief Psychiatric Rating Scale - Extended (BPRS+)
   * Life Satisfaction Scale (LS)
   * Positive and Negative Affect Schedule (PANAS)
   * Harmony in Life Scale (HILS)
   * Ten Item Personality Inventory (TIPI)
   * Honesty-Humility Scale (HH)

   Extended Follow-Up Phase (Week 24-52) 9-Month Follow-Up (Week 36)
   * Eating Disorder Examination Questionnaire (EDE-Q )
   * Columbia-Suicide Severity Rating Scale (C-SSRS)
   * Brief Psychiatric Rating Scale - Extended (BPRS+)
   * AE/SAE monitoring
   * BMI, blood pressure, ECG
   * Fasting glucose, U-tox

     12-Month Final Follow-Up (Week 52)
   * Eating Disorder Examination Questionnaire (EDE-Q )
   * Columbia-Suicide Severity Rating Scale (C-SSRS)
   * Brief Psychiatric Rating Scale - Extended (BPRS+)
   * Patient Health Questionnaire (PHQ-9)
   * Generalized Anxiety Disorder scale (GAD-7)
   * Ten Item Personality Inventory (TIPI)
   * Meaningful Life Experience Rating (MLE).
   * AE/SAE monitoring
   * BMI, blood pressure, ECG
   * Fasting glucose, U-tox Participants who show signs of psychological or physical deterioration at any point during the study between follow-ups are instructed to contact the research team at any time and will be offered additional assessment and support.

   Description of Psilocybin Administration and Psychological support Psychological support includes a non-directive preparation and integration pre- and post-dosing sessions according to protocol manual, alongside support for the patient on the dosing session day. The study follows the guidelines for safe research with psychedelics. Preparation session will include psychoeducation of the effects of psilocybin, breathing techniques, getting to know the two therapists (one male and one female). A standardized preparation script will ensure consistency across participants. The two integration sessions following each dosing session last 1-2 h and focus on exploring the session's effects and offer support in integrating the experience. Integration sessions will include structured discussions about insights gained, with therapists facilitating connections between the experience and the participant's therapeutic goals. The therapists will be licensed healthcare professionals.

   Dosing session day The dosing session, lasting 6-8 hours, is supported by the therapists introduced during preparation sessions. The psilocybin's acute effects persist for 4-6 hours, recorded via video and audio. Participants, lie down with an optional eye mask, experience the session in a comfortable room with a pre-selected music playlist, respecting individual preferences. Therapists provide support and guidance if requested but with minimal psychotherapeutic focus. Therapists will follow pre-established protocols for de-escalation and grounding in case of distressing experiences. Parents are introduced at the session's end with participant approval. During the dosing session, a medically trained study doctor will be available, equipped for emergencies in the unlikely event of serious adverse events related to psilocybin risks.

   Biological Sampling Procedures Blood samples will be collected for the analysis of Brain-Derived Neurotrophic Factor (BDNF) as the primary biomarker and for tolerance and safety measurements. Additionally, we aim to collect one tube of additional whole blood per occasion for future analysis.

   BDNF samples will be taken at five key time points: (1) before treatment (baseline), (2) and (3) at first integration session after Psilocybin 25mg dosing, (4) at 8 weeks, and (5) during the 6-month follow-up. This ensures comprehensive longitudinal data collection.

   Blood samples of glucose, kidney and liver status will be measured at the same time points as above for safety and tolerance reasons. None of these blood samples are collected or stored.

   All blood samples are done by a standard peripheral venous sampling method performed by a nurse at the research facility at the university hospital clinic for psychiatry at Baravägen 1, Lund.

   Procedures will be implemented to minimize discomfort during blood collection, such as using pediatric needles for younger participants when necessary. Blood collection and processing will follow standardized protocols to ensure sample integrity.

   Discontinuation from the Clinical Trial

   A participant will be discontinued entirely from the clinical trial (i.e., all further participation and follow-up will end) only under the following condition:

   Withdrawal of informed consent at any time, for any reason, without the need to justify.

   Discontinuation from the Intervention (Dosing) Participants may be discontinued from the intervention (i.e., psilocybin administration - first or second dose), without being excluded from the trial. Participants will be encouraged to continue with follow-up assessments unless they explicitly withdraw consent. This approach allows for continued safety and data collection in accordance with the intention-to-treat principle.

   Reasons for discontinuing intervention may include:
   * Development or discovery of exclusion criteria after inclusion (e.g. new psychiatric diagnosis, pregnancy).
   * Emergence of a serious adverse event (SAE) or medical condition that, in the investigator's judgment, makes continued treatment unsafe.
   * Initiation of treatment with prohibited medication according to protocol.
   * Failure to adhere to critical aspects of the study protocol (e.g. repeated missed visits, non-compliance with preparation or safety procedures).
   * Investigator decision in consultation with the medical monitor.

   The reason for discontinuation will be documented. Participants will be offered a final follow-up visit when appropriate.

   Non-compliance to fMRI will not lead to study exclusion nor discontinuation of the intervention.

   Methods for Measurement of Endpoints for Clinical Safety Continuous clinical safety monitoring will be performed by licensed healthcare professionals at Lund University Hospital throughout the trial, from baseline to the final 12-month follow-up. The safety evaluations cover physical, biochemical, and psychological parameters relevant to psilocybin administration.

   Measurements for assessing clinical safety will include blood samples of hepatic and renal function, glucose, urine toxicology, cardiovascular parameters, assessment of suicidality, assessment of mental health symptoms and and assessment of Adverse Events/Serious Adverse Events/Suspected Unexpected Serious Adverse Reactions (AE/SAE/SUSARs).

   Assessment of Adverse Events Participants are instructed to contact the research team during daytime hours for urgent concerns. Outside of study hours, they are directed to seek emergency services. Events will be assessed by the clinical team for causality, intensity, and seriousness and potential relationship to treatment (psilocybin 25mg).

   The investigator is responsible for determining whether there is a causal relationship between the AE/SAE and use of the investigational medicinal product.

   Consideration should be given to whether there is a reasonable possibility of establishing a causal relationship between the adverse event and the investigational medicinal product based on the analysis of the available evidence.

   All AE can be categorized as either likely related, possibly related, unlikely related or not related.

   Those AEs which are suspected of having a causal relationship to the investigational medicinal product will be followed up until the subject has recovered or is well taken care of and on the way to good recovery. Each adverse event shall be classified by an investigator as mild, moderate or severe.

   Follow-up of Adverse Events Follow-up visits will be scheduled for all participants experiencing AEs to ensure resolution and ongoing safety.

   Participants with unresolved AEs at the end of the trial will be monitored until resolution or stabilization.

   For SAEs, additional follow-ups will be scheduled at least every two weeks until resolution. The frequency can be changed by the Safety Review Committee or Principal Investigator.

   Procedures in Case of Emergencies and Overdose Emergency protocols are in place, including immediate medical care and monitoring.

   In case of an overdose, the participant will be transferred to an emergency facility. Emergency kits, including benzodiazepines for anxiety or seizures, will be available during all dosing sessions.

   Pregnancy Management Participants who can become pregnant must use a highly effective form of contraception during the study and for two months after the last psilocybin dose. Approved methods include hormonal contraception, IUDs, sterilization, vasectomized partner, or abstinence. Urine pregnancy tests will be done at screening, before each psilocybin session, and as needed during follow-up. Psilocybin's effects on pregnancy are unknown. To reduce possible risks, strict contraception and testing protocols are required.

   Interim Analysis Following two administration sessions of 25mg psilocybin, a panel of three senior psychiatrists, who are not part of the research team, will conduct an evaluation of the safety data and adherence to the protocol. This analysis will be repeated after a total of 20 psilocybin administrations have been completed. After 25 patients over 18 have been through dosing sessions, patients 16-17 will be recruited.

   Methods for Measurement of Endpoints for Clinical Efficacy

   Composite Relapse Endpoint:

   BMI Decrease: Measured at baseline, 8 weeks, and 6 months using calibrated equipment and standardized protocols.

   Hospitalization Data: Collected through patient reports and confirmed by medical records.

   Symptom Deterioration: Assessed using validated tools such as the EDE-Q 6.0 and clinical interviews conducted by trained staff.

   Clinical Intervention Use: Recorded in patient files, including initiation of new treatments during follow-up.

   Statistics Analysis Population Both the Intention-to-treat (ITT) and per-protocol populations will be analyzed.

   ITT analysis will include all participants who are randomized, regardless of protocol adherence, to ensure generalizability. Per-protocol analysis will focus on participants who completed the study as planned, ensuring the assessment of efficacy under ideal conditions.

   Statistical Analyses

   Primary Baseline Analyses:

   The primary analyses will involve descriptive statistics for demographic and baseline characteristics, ensuring comparability across groups, and control for follow-up measurements.

   Primary Endpoints analysis We will analyze differences in the number of participants and severity experiencing adverse event/serious adverse event (AE/SAE) between the groups standardized forms for AE/SAE capturing: Event description, Start and end dates, Severity (e.g., mild, moderate, severe), Relatedness to intervention (assessed by safety review committee), Action taken.

   The primary statistical methods will be:

   Descriptive Frequencies and Percentages. Comparing Proportions (Most Common for "Incidence") (Chi-squared test (or Fisher's Exact Test): Fisher's exact test is preferred for small cell counts (<5).

   Risk Ratio (RR) or Odds Ratio (OR) with Confidence Intervals: Report these measures of effect size to quantify the magnitude and precision of the difference between groups. An RR > 1 would indicate a higher risk in the intervention group.

   Comparing Severity and Relatedness is assessed with Mann-Whitney U test or Student t-test to compare severity distributions between groups.

   Secondary Endpoints:

   For secondary endpoints (e.g., changes in fMRI connectivity, BDNF, rating scales), group comparisons, including t-test, Analysis of Variance (ANOVA), and Repeated Measures ANOVA will be utilized. When controlling for variables such as individual differences, ANCOVA or Multivariate Analysis of Covariance (MANCOVA) will be utilized. Principal component analysis (PCA) or independent component analysis (ICA) may be applied to identify patterns in fMRI data. Endpoints include longitudinal between- and within-person analyses.

   When dichotomous (binary) outcome variables: Binary outcomes (e.g., remission, response rates) will be analyzed using logistic regression models, adjusting for baseline characteristics such as age, baseline BMI, and symptom severity. The odds ratios and 95% confidence intervals will be reported.

   When continuous (dimensional) variables (e.g., BMI, BDNF levels, cognitive flexibility) will be analyzed using linear mixed-effects models, and regression models of various types.

   Other: Exploratory Subgroup Analyses:

   Exploratory subgroup analyses will assess treatment effects across different strata (e.g., age groups, baseline severity) using interaction terms in regression models or stratified analyses to explore heterogeneity in treatment responses.

   Other: Sensitivity Analyses:

   Sensitivity analyses will address missing data using methods such as multiple imputation or maximum likelihood estimation. These methods ensure robustness of the findings by accounting for the potential impact of missing data on primary and secondary outcomes.

   Adjustment of Significance and Confidence Interval A Bonferroni correction or false discovery rate (FDR) adjustment will be applied for multiple comparisons to control Type I error.

   Results will be presented with 95% confidence intervals, and significance will be set at a two-tailed p-value of <0.05 after adjustments.

   Ethical considerations This research aims to address the urgent clinical need presented by anorexia nervosa, a condition with alarmingly high mortality rates and no effective pharmacological treatments, while maintaining the highest ethical standards. Psilocybin has shown potential in addressing treatment-resistant conditions across other psychiatric diagnoses. Through comprehensive safety measures, informed consent, and support tailored to participants' needs, the study seeks to minimize risks and contribute valuable insights into both anorexia nervosa treatment and the broader therapeutic potential of psilocybin.

   Previous research using doses of 30 and 40 mg reported no serious adverse events. Key risks of psilocybin, as noted in literature, include prolonged psychotic symptoms, flashback phenomena or Hallucinogen Persisting Perceptual Disorder (HPPD), and anxiety reactions. Studies at the John Hopkins Center for Psychedelic Research, encompassing over 300 participants and 600 dosing sessions with 25mg psilocybin, recorded no cases of HPPD. HPPD itself is rare, with a prevalence of 4-4.5% among lifetime users of hallucinogens, though the specific incidence related to psilocybin is unclear. Prolonged psychotic responses in clinical psilocybin studies are infrequent, less than 1%. Anxiety during psilocybin experiences is common. A survey involving 1993 participants (mean age 29) exploring challenging experiences with psilocybin found that 84% benefited, despite psychological distress. The severity of the experience positively correlated with long-term increases in well-being. This study includes robust preparatory and integration sessions to minimize distress and maximize therapeutic outcomes. Therapists will receive specialized training to handle challenging experiences in real time.

   Although the MRI examinations, during which patients need to lie still for about 1 hour, might be perceived as uncomfortable by some, they pose no health risk for the patient if routine safety precautions are followed (i.e. careful screening for contraindications for undergoing MRI and ensuring that no ferromagnetic metal objects are brought near the scanner).

   Specific clinical AN related risk One study of psilocybin 25mg for adults with AN, reported no clinically significant changes in ECG, vital signs, or suicidality levels. Only two participants experienced asymptomatic hypoglycemia post-treatment, which resolved within 24 hours. Additionally, no significant changes were noted in laboratory values. All adverse events (AEs) observed were mild and temporary. The overall participant feedback indicated that the treatment was generally well-received and deemed acceptable. To mitigate potential risks, participants in this study will undergo comprehensive medical screening, including blood tests and ECG, before dosing session. A trained physician will be available during all psilocybin sessions to address medical emergencies, if needed.

   Suicidality and psilocybin A study on psilocybin for depression treatment noted two cases of suicidal behavior in the 25 mg group, compared to two in the 10 mg group and none in the 1 mg group within three weeks post-dosing. Another study comparing 25mg psilocybin with escitalopram for depression found no increase in serious adverse events or suicidal behavior in either group. This study includes active monitoring for suicidal ideation and behaviour during and after treatment sessions, with immediate intervention plans in place.

   Procedure for Obtaining Informed Consent Informed consent will be obtained from all participants, including both parents or other caregiver when patient is between 16-17. Participants will receive detailed written and verbal information about the trial's purpose, procedures, potential risks, and benefits. They will have the opportunity to ask questions and consult with family members or advisors before consenting. Care will be taken to ensure that minors understand the study in an age-appropriate manner. A cooling-off period of at least 48 hours will be provided between the provision of information and consent signing to allow participants to make an informed decision.

   Data Protection Data will be pseudonymized and handled according to GDPR. Only study personnel with relevant clearance will have access to identifiable data. Pseudonymized data will be stored securely on encrypted servers. A data management plan will outline the procedures for data collection, storage, sharing, and destruction, ensuring compliance with GDPR and ethical standards. Informed consent will include explicit information about data handling, potential use in future research, and participants' right to withdraw consent for data use at any time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AN per DSM-5
* Have experienced at least one period of remission (minimum BMI 17) followed by a relapse
* Age 16-35
* BMI >16
* Stable contact with a psychiatric unit
* Ability to provide informed consent

Exclusion Criteria:

* Psychosis, bipolar disorder, substance use disorder, family history of psychosis or bipolar disorder, refusal of birth control, lifetime psychedelic use, unable to washout ongoing medications* that would interfere negatively with the study drug
* Cardiovascular conditions
* Resting systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg at screening or baseline
* Clinically significant arrhythmias, tachycardia and QT prolongation
* History of stroke, myocardial infarction, or other significant cardiovascular events
* Seizure disorders or history of epilepsy
* Diabetes mellitus, positive drug tests, suicidal intent, allergy or intolerance to drug content, blood or needle phobia
* Only for the MRI-part of the study: Metal pieces in the body (contraindicated by fMRI, assessed in each case by MR-technician). Non-compliance to fMRI will not lead to study exclusion
* Any other clinically significant medical condition that, in the investigator's opinion, may pose a risk to the participant or interfere with study results
* Care under the Swedish Compulsory Psychiatric Care Act (LPT)

  * 5-HT2A-antagonist need two weeks washout

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of psilocybin 25 mg in young adults with anorexia nervosa, as measured by incidence of adverse events (AEs) and serious adverse events (SAEs). | From enrollment to the end of trial 12 month post-baseline.
  Adverse events (AEs) refers to any unwelcome medical occurrence in a patient who has been administered psilocybin or TAU, which may not necessarily be caused by the treatment. Serious Adverse Event (SAE) includes any medical incident or effect, irrespective of dosage, that a) leads to death, b) is life-threatening, c) necessitates hospitalization, or d) results in persistent or significant disability or incapacity.
  Events will be assessed by the clinical team for causality, intensity, and seriousness and potential relationship to treatment (psilocybin or TAU). All AEs will be categorized based on their severity and likelihood of treatment attribution.

SECONDARY OUTCOMES:
To evaluate the efficacy of two doses of psilocybin, administred with psychological support, in reducing AN symptoms compared to TAU, as measured by time to response, time to remission and time to relapse. | Efficacy will be evaluated during the 12-month follow-up.
  Response defined as a significant improvement in weight and psychological symptoms: 1) BMI Increase: ≥10% increase in BMI from baseline or 2) reaching a BMI ≥18.5 if achievable within the study period.
  Remission defined as achieving and maintaining weight restoration and psychological well-being, with no significant symptoms of anorexia nervosa:
  1) Weight Restoration of BMI ≥18.5 sustained for at least four weeks, or 2) a weight within 90-95% of ideal body weight adjusted for age and height.
  Relapse defined as: 1) ≥7 % decrease in BMI compared to post-hospitalization baseline BMI; 2) Re-hospitalization for anorexia nervosa-related complications; 3) Initiation of additional intensive psychiatric or nutritional interventions, including day-patient or inpatient programs; or 4) Self-reported significant deterioration in eating disorder symptoms as assessed by validated scales such as the Eating Disorder Examination Questionnaire 6.0.
Assess potential mechanisms of action through neuroimaging (fMRI), before and after the two-dose psilocybin treatment, administered with psychological support | fMRI will be preformed at baseline (week 0), after first dosing (week 1) and at primary endpoint (week 8).
  Investigate potential mechanisms of action, i.e. change in brain resting state connectivity, as measured by fMRI, before and after the two-dose psilocybin treatment, administered with psychological support
Changes in serum brain-derived neurotrophic factor (BDNF) levels from before and after treatment with two doses of 25 mg psilocybin, administered with psychological support. | BDNF will be measured at baseline (week 0), after second dosing (week 4), at primary end point (week 8) and at 6-month follow-up
  Serum BDNF will be measured in blood samples to investigate potential mechanisms of action.
To conduct a qualitative analysis of how participants, their relatives, and therapists experience and perceive the intervention | Assessments will be preformed at different timepoints during the 12-month follow-up.
  Qualitative analysis will be done based on semi-structured interviews, investigating the experience of the intervention from the above mentioned parts. Data will be analyzed thematically to identify common themes and patterns across participants' reports.
To assess changes in symtoms of depression before and after two-doses of psilocybin, administered with psychological support, in young adults with anorexia nervosa. | Changes will be assessed at baseline and then repeatedly within the 12-month follow-up
  Symtoms of depression will be assessed by ussing PHQ-9 (Patient Health Questionnaire-9). PHQ-9 is a self-report instrument with 9 items assessing depressive symptoms over the past two weeks. Each item is scored from 0 (not at all) to 3 (nearly every day), giving a total score ranging from 0 to 27. Higher scores indicate greater severity of depressive symptoms. The outcome is defined as the change in total PHQ-9 score.
To assess changes in symtoms of anxiety before and after two-doses of psilocybin, administered with psychological support, in young adults with anorexia nervosa. | Changes will be assessed at baseline and then repeatedly within the 12-month follow-up.
  Symtoms of anxiety will be assessed by using the GAD-7 (Generalized Anxiety Disorder-7). GAD-7 is a self-report questionnaire with 7 items assessing anxiety symptoms over the past two weeks. Each item is scored from 0 (not at all) to 3 (nearly daily), resulting in a total score ranging from 0 to 21. Higher scores indicate greater severity of anxiety symptoms.
To assess changes in eating disorder symptoms before and after two-doses of psilocybin, administered with psychological support, in young adults with anorexia nervosa. | Changes will be assessed at baseline and then repeatedly within the 12-month follow-up.
  Change in eating disorder symtoms will be assessed by using the EDE-Q 6.0 (Eating Disorder Examination Questionnaire 6.0). EDE-Q 6.0 is a self-report instrument assessing the range and severity of eating disorder symptoms over the past 28 days. It contains 28 items that gives four subscale scores, each scored from 0 to 6, with higher scores indicating greater symptom severity. A Global Score is calculated as the mean of the four subscale scores. Items are rated on a 7-point scale ranging from 0 (no days) to 6 (every day). The Global Score ranges from 0.0 to 6.0, with higher scores indicating greater symptom severity.
To assess changes in suicidal ideation and behavior before and after two-doses of psilocybin, administered with psychological support, in young adults with anorexia nervosa. | Changes will be assessed at baseline and then repeatedly within the 12-month follow-up.
  Changes in suicidal ideation and behavior will be assessed using the Columbia-Suicide Severity Rating Scale (C-SSRS) which is a structured instrument to assess the severity and intensity of suicidal ideation and behavior. The scale evaluates the presence of suicidal thoughts, the intensity of ideation and any suicidal or self-injurious behaviors. Suicidal ideation severity is rated on a 5-point ordinal scale (1 = wish to be dead to 5 = suicidal intent with plan). Higher scores indicate greater severity of suicidal ideation. Suicidal behavior is recorded as present/absent for different type.
To assess changes in psychiatric symptom severity before and after two-doses of psilocybin, administered with psychological support, in young adults with anorexia nervosa. | Changes will be assessed at baseline and then repeatedly within the 12-month follow-up.
  The Brief Psychiatric Rating Scale - Extended (BPRS+) will be used to assess change in a broad range of psychiatric symptoms, including positive symptoms, negative symptoms and affective symptoms. The BPRS+ consists of 24 items, each rated on a 7-point Likert scale from 1 (not present) to 7 (extremely severe). Total scores are obtained by summing all items, yielding a range from 24 to 168. Higher scores indicate greater overall symptom severity.
To assess changes in life satisfaction before and after two-doses of psilocybin, administered with psychological support, in young adults with anorexia nervosa. | Changes will be assessed at baseline and then repeatedly within the 6-month follow-up.
  The Life Satisfaction Scale (LS) is a self-report instrument designed to assess overall satisfaction with life, this scale will be used to assess change in life satisfaction. Respondents rate items on a scale (commonly 1 = strongly disagree to 7 = strongly agree). A total score is calculated by summing item scores of the 5 items, giving a total score between 5 to 35. Higher scores indicate greater overall life satisfaction.
To assess changes in positive and negative affect before and after two-doses of psilocybin, administered with psychological support, in young adults with anorexia nervosa. | Changes will be assessed at baseline and then repeatedly within the 6-month follow-up.
  The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire that assesses two dimensions of mood: Positive Affect (PA) and Negative Affect (NA). PANAS will be used to assess change in positive and negative affect. The standard PANAS consists of 20 items, with 10 items for PA and 10 items for NA. Each item is rated on a 5-point scale ranging from 1 (very slightly or not at all) to 5 (extremely). Subscale scores are calculated by summing responses, giving a range of 10 to 50 for each subscale. Higher PA scores indicate greater positive affect, while higher NA scores indicate greater negative affect.
To assess changes in harmony in life before and after two-doses of psilocybin, administered with psychological support, in young adults with anorexia nervosa. | Changes will be assessed at baseline and then repeatedly within the 6-month follow-up.
  The Harmony in Life Scale (HILS) is a self-report measure designed to assess perceived sense of balance, congruence, and harmony in their lives. The scale consists of 5 items, each rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). A total score is calculated as the mean of the items, with possible scores ranging from 1.0 to 7.0. Higher scores indicate a greater perceived harmony in life.
To assess changes in personality traits before and after two-doses of psilocybin, administered with psychological support, in young adults with anorexia nervosa. | Changes will be assessed at baseline and then repeatedly within the 12-month follow-up.
  Changes in personality traits will be assessed using the Ten Item Personality Inventory (TIPI). TIPI is a self-report instrument designed to assess the Big Five personality dimensions. It consists of 10 items, with 2 items per trait. Each item is rated on a 7-point scale ranging from 1 (disagree strongly) to 7 (agree strongly). Scores for each trait are calculated as the mean of the 2 relevant items, giving a range from 1.0 to 7.0. Higher scores indicate greater expression of the respective personality trait.
Change in dark personality traits measured by the Honesty-Humility Scale (HH) before and after two psilocybin dosing sessions with psychological support in young adults with anorexia nervosa | Changes will be assessed at baseline and then repeatedly within the 6-month follow-up.
  Change in dark personality traits will be assessed using the Honesty-Humility (HH) scale, a self-report subscale of the HEXACO personality inventory. The HH scale includes items covering four facets: sincerity, fairness, greed avoidance, and modesty. The outcome is defined as the change in HH scores before and after two psilocybin dosing sessions with psychological support.
To assess how treatment expectation affect outcomes of two-doses of psilocybin, administered with psychological support, in young adults with anorexia nervosa. | Treatment expectations will be measured at baseline with the Expectation for Treatment Scale - Brief Form (ETS-BF).
  The Expectation for Treatment Scale - Brief Form (ETS-BF) is a self-report instrument with 5 items that assess expectations regarding treatment outcomes. Each item is rated on a 4-point scale, ranging from 1 (partially disagree) to 4 (definitely agree). Scores are summed to produce a total score ranging from 5 to 20, with higher scores reflecting greater positive expectations of treatment effectiveness.
Readiness and motivation for change assessed by the RMQ before and after two psilocybin doses with psychological support in young adults with anorexia nervosa | Changes will be assessed at baseline and then repeatedly within the 6-month follow-up.
  The Readiness and Motivation Questionnaire (RMQ) is a self-report instrument designed to assess readiness for change in eating disorder symptoms. It evaluates four symptom domains and provides four subscale scores within each domain. Items are rated on a scale, and subscale scores are calculated separately for each domain and dimension. The questionnaire is not designed to produce a single overall total score, instead it provides a profile of readiness across domains and subscales.
To assess changes in general change mechanisms before and after two-doses of psilocybin, administered with psychological support, in young adults with anorexia nervosa. | Changes will be assessed at baseline and then repeatedly within the 6-month follow-up.
  The General Change Mechanisms Questionnaire (GCMQ) is a self-report instrument developed to assess five empirically established common therapeutic change mechanisms within the context of psychedelic experiences. This questionnaire will be used to assess participants' experiences of therapeutic change mechanisms before and after treatment. Scores are calculated separately for each mechanism, and higher scores indicate stronger endorsement of that particular change process.

CONTACTS AND LOCATIONS:
Overall Officials: Pouya Movahed Rad, Associate Professor, Principal Investigator — Department of Clinical Sciences, Lund University, Sweden
Locations (1):
- Psykiatrikliniken, Baravägen 1, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carhart-Harris R, Giribaldi B, Watts R, Baker-Jones M, Murphy-Beiner A, Murphy R, Martell J, Blemings A, Erritzoe D, Nutt DJ. Trial of Psilocybin versus Escitalopram for Depression. N Engl J Med. 2021 Apr 15;384(15):1402-1411. doi: 10.1056/NEJMoa2032994. PMID 33852780
- [Background] Goodwin GM, Aaronson ST, Alvarez O, Arden PC, Baker A, Bennett JC, Bird C, Blom RE, Brennan C, Brusch D, Burke L, Campbell-Coker K, Carhart-Harris R, Cattell J, Daniel A, DeBattista C, Dunlop BW, Eisen K, Feifel D, Forbes M, Haumann HM, Hellerstein DJ, Hoppe AI, Husain MI, Jelen LA, Kamphuis J, Kawasaki J, Kelly JR, Key RE, Kishon R, Knatz Peck S, Knight G, Koolen MHB, Lean M, Licht RW, Maples-Keller JL, Mars J, Marwood L, McElhiney MC, Miller TL, Mirow A, Mistry S, Mletzko-Crowe T, Modlin LN, Nielsen RE, Nielson EM, Offerhaus SR, O'Keane V, Palenicek T, Printz D, Rademaker MC, van Reemst A, Reinholdt F, Repantis D, Rucker J, Rudow S, Ruffell S, Rush AJ, Schoevers RA, Seynaeve M, Shao S, Soares JC, Somers M, Stansfield SC, Sterling D, Strockis A, Tsai J, Visser L, Wahba M, Williams S, Young AH, Ywema P, Zisook S, Malievskaia E. Single-Dose Psilocybin for a Treatment-Resistant Episode of Major Depression. N Engl J Med. 2022 Nov 3;387(18):1637-1648. doi: 10.1056/NEJMoa2206443. PMID 36322843
- [Background] Carbonaro TM, Bradstreet MP, Barrett FS, MacLean KA, Jesse R, Johnson MW, Griffiths RR. Survey study of challenging experiences after ingesting psilocybin mushrooms: Acute and enduring positive and negative consequences. J Psychopharmacol. 2016 Dec;30(12):1268-1278. doi: 10.1177/0269881116662634. Epub 2016 Aug 30. PMID 27578767
- [Background] Carhart-Harris RL, Bolstridge M, Rucker J, Day CM, Erritzoe D, Kaelen M, Bloomfield M, Rickard JA, Forbes B, Feilding A, Taylor D, Pilling S, Curran VH, Nutt DJ. Psilocybin with psychological support for treatment-resistant depression: an open-label feasibility study. Lancet Psychiatry. 2016 Jul;3(7):619-27. doi: 10.1016/S2215-0366(16)30065-7. Epub 2016 May 17. PMID 27210031
- [Background] Studerus E, Kometer M, Hasler F, Vollenweider FX. Acute, subacute and long-term subjective effects of psilocybin in healthy humans: a pooled analysis of experimental studies. J Psychopharmacol. 2011 Nov;25(11):1434-52. doi: 10.1177/0269881110382466. Epub 2010 Sep 20. PMID 20855349
- [Background] Kurtom M, Henning A, Espiridion ED. Hallucinogen-persisting Perception Disorder in a 21-year-old Man. Cureus. 2019 Feb 14;11(2):e4077. doi: 10.7759/cureus.4077. PMID 31019855
- [Background] Bogenschutz MP, Ross S, Bhatt S, Baron T, Forcehimes AA, Laska E, Mennenga SE, O'Donnell K, Owens LT, Podrebarac S, Rotrosen J, Tonigan JS, Worth L. Percentage of Heavy Drinking Days Following Psilocybin-Assisted Psychotherapy vs Placebo in the Treatment of Adult Patients With Alcohol Use Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Oct 1;79(10):953-962. doi: 10.1001/jamapsychiatry.2022.2096. PMID 36001306
- [Background] Griffiths RR, Johnson MW, Richards WA, Richards BD, McCann U, Jesse R. Psilocybin occasioned mystical-type experiences: immediate and persisting dose-related effects. Psychopharmacology (Berl). 2011 Dec;218(4):649-65. doi: 10.1007/s00213-011-2358-5. Epub 2011 Jun 15. PMID 21674151
- [Background] Griffiths RR, Richards WA, McCann U, Jesse R. Psilocybin can occasion mystical-type experiences having substantial and sustained personal meaning and spiritual significance. Psychopharmacology (Berl). 2006 Aug;187(3):268-83; discussion 284-92. doi: 10.1007/s00213-006-0457-5. Epub 2006 Jul 7. PMID 16826400
- [Background] Johnson M, Richards W, Griffiths R. Human hallucinogen research: guidelines for safety. J Psychopharmacol. 2008 Aug;22(6):603-20. doi: 10.1177/0269881108093587. Epub 2008 Jul 1. PMID 18593734
- [Background] Nakazato M, Hashimoto K, Shimizu E, Kumakiri C, Koizumi H, Okamura N, Mitsumori M, Komatsu N, Iyo M. Decreased levels of serum brain-derived neurotrophic factor in female patients with eating disorders. Biol Psychiatry. 2003 Aug 15;54(4):485-90. doi: 10.1016/s0006-3223(02)01746-8. PMID 12915293
- [Background] Ly C, Greb AC, Cameron LP, Wong JM, Barragan EV, Wilson PC, Burbach KF, Soltanzadeh Zarandi S, Sood A, Paddy MR, Duim WC, Dennis MY, McAllister AK, Ori-McKenney KM, Gray JA, Olson DE. Psychedelics Promote Structural and Functional Neural Plasticity. Cell Rep. 2018 Jun 12;23(11):3170-3182. doi: 10.1016/j.celrep.2018.05.022. PMID 29898390
- [Background] Cohen-Cory S, Kidane AH, Shirkey NJ, Marshak S. Brain-derived neurotrophic factor and the development of structural neuronal connectivity. Dev Neurobiol. 2010 Apr;70(5):271-88. doi: 10.1002/dneu.20774. PMID 20186709
- [Background] Lohof AM, Ip NY, Poo MM. Potentiation of developing neuromuscular synapses by the neurotrophins NT-3 and BDNF. Nature. 1993 May 27;363(6427):350-3. doi: 10.1038/363350a0. PMID 8497318
- [Background] Siegel JS, Subramanian S, Perry D, Kay B, Gordon E, Laumann T, Reneau R, Gratton C, Horan C, Metcalf N, Chacko R, Schweiger J, Wong D, Bender D, Padawer-Curry J, Raison C, Raichle M, Lenze EJ, Snyder AZ, Dosenbach NUF, Nicol G. Psilocybin desynchronizes brain networks. medRxiv [Preprint]. 2023 Aug 24:2023.08.22.23294131. doi: 10.1101/2023.08.22.23294131. PMID 37701731
- [Background] Daws RE, Timmermann C, Giribaldi B, Sexton JD, Wall MB, Erritzoe D, Roseman L, Nutt D, Carhart-Harris R. Increased global integration in the brain after psilocybin therapy for depression. Nat Med. 2022 Apr;28(4):844-851. doi: 10.1038/s41591-022-01744-z. Epub 2022 Apr 11. PMID 35411074
- [Background] Peck SK, Shao S, Gruen T, Yang K, Babakanian A, Trim J, Finn DM, Kaye WH. Psilocybin therapy for females with anorexia nervosa: a phase 1, open-label feasibility study. Nat Med. 2023 Aug;29(8):1947-1953. doi: 10.1038/s41591-023-02455-9. Epub 2023 Jul 24. PMID 37488291
- [Background] Foldi CJ, Liknaitzky P, Williams M, Oldfield BJ. Rethinking Therapeutic Strategies for Anorexia Nervosa: Insights From Psychedelic Medicine and Animal Models. Front Neurosci. 2020 Feb 4;14:43. doi: 10.3389/fnins.2020.00043. eCollection 2020. PMID 32116500
- [Background] MacLean KA, Johnson MW, Griffiths RR. Mystical experiences occasioned by the hallucinogen psilocybin lead to increases in the personality domain of openness. J Psychopharmacol. 2011 Nov;25(11):1453-61. doi: 10.1177/0269881111420188. Epub 2011 Sep 28. PMID 21956378
- [Background] Carhart-Harris RL, Goodwin GM. The Therapeutic Potential of Psychedelic Drugs: Past, Present, and Future. Neuropsychopharmacology. 2017 Oct;42(11):2105-2113. doi: 10.1038/npp.2017.84. Epub 2017 Apr 26. PMID 28443617
- [Background] Mertens LJ, Preller KH. Classical Psychedelics as Therapeutics in Psychiatry - Current Clinical Evidence and Potential Therapeutic Mechanisms in Substance Use and Mood Disorders. Pharmacopsychiatry. 2021 Jul;54(4):176-190. doi: 10.1055/a-1341-1907. Epub 2021 Jan 20. PMID 33472250
- [Background] Swanson LR. Unifying Theories of Psychedelic Drug Effects. Front Pharmacol. 2018 Mar 2;9:172. doi: 10.3389/fphar.2018.00172. eCollection 2018. PMID 29568270
- [Background] Halmi KA, Goldberg SC, Casper RC, Eckert ED, Davis JM. Pretreatment predictors of outcome in anorexia nervosa. Br J Psychiatry. 1979 Jan;134:71-8. doi: 10.1192/bjp.134.1.71. PMID 760925
- [Background] Halmi KA. Perplexities of treatment resistance in eating disorders. BMC Psychiatry. 2013 Nov 7;13:292. doi: 10.1186/1471-244X-13-292. PMID 24199597
- [Background] Khalsa SS, Portnoff LC, McCurdy-McKinnon D, Feusner JD. What happens after treatment? A systematic review of relapse, remission, and recovery in anorexia nervosa. J Eat Disord. 2017 Jun 14;5:20. doi: 10.1186/s40337-017-0145-3. eCollection 2017. PMID 28630708
- [Background] Steinhausen HC. The outcome of anorexia nervosa in the 20th century. Am J Psychiatry. 2002 Aug;159(8):1284-93. doi: 10.1176/appi.ajp.159.8.1284. PMID 12153817
- [Background] DeJong H, Oldershaw A, Sternheim L, Samarawickrema N, Kenyon MD, Broadbent H, Lavender A, Startup H, Treasure J, Schmidt U. Quality of life in anorexia nervosa, bulimia nervosa and eating disorder not-otherwise-specified. J Eat Disord. 2013 Nov 26;1:43. doi: 10.1186/2050-2974-1-43. eCollection 2013. PMID 24999421
- [Background] Westmoreland P, Krantz MJ, Mehler PS. Medical Complications of Anorexia Nervosa and Bulimia. Am J Med. 2016 Jan;129(1):30-7. doi: 10.1016/j.amjmed.2015.06.031. Epub 2015 Jul 10. PMID 26169883
- [Background] Arcelus J, Mitchell AJ, Wales J, Nielsen S. Mortality rates in patients with anorexia nervosa and other eating disorders. A meta-analysis of 36 studies. Arch Gen Psychiatry. 2011 Jul;68(7):724-31. doi: 10.1001/archgenpsychiatry.2011.74. PMID 21727255